CLINICAL TRIAL: NCT04042077
Title: A Randomized, Observer-blinded, Active-controlled, Phase Illb Study to Compare IV / Oral Delafloxacin Fixed-dose Monotherapy With Best Available Treatments in a Microbiologically Enriched Population With Surgical Site Infections
Brief Title: Delafloxacin IV and OS Administration Compared to Best Available Therapy in Patients With Surgical Site Infections
Acronym: DRESS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: COVID-19 seriously affected the study execution as required by the protocol
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DELA-01; 2018-001082-17 (EudraCT Number)
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Results first posted 2021-10-29 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2020-11

CONDITIONS: Surgical Site Infection
Keywords: Infection, Surgical Infection
MeSH Terms: conditions — Surgical Wound Infection; Infections | interventions — delafloxacin; Vancomycin; Linezolid; Piperacillin, Tazobactam Drug Combination; Tigecycline

STUDY DESIGN:
Intervention Model Description: The study will compare delafloxacin against best available therapy selected by the investigator for the cardiothoracic/leg related or abdominal site infection
Who Masked: Outcomes Assessor
Masking Description: Only the blinded observer will be unaware of the treatment assigned to patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Delafloxacin (Experimental): Delafloxacin IV, with the option to switch to delafloxacin oral
  Interventions: Drug: Delafloxacin
- Best Available Therapy (Active Comparator): Cardiothoracic / related leg SSI
  * Vancomycin IV
  * Linezolid IV, with the option to switch to linezolid oral.
  In case of suspicion of Gram-negative, additional therapy shall be added as per investigator's choice
  Abdominal SSI
  * Piperacillin/Tazobactam IV, OR
  * Tigecycline IV
  In case of suspicion of MRSA, if the pre-selected treatment is Piperacillin/Tazobactam, additional therapy shall be added as per investigator's choice.
  Interventions: Drug: Vancomycin; Drug: Linezolid; Drug: Piperacillin/Tazobactam; Drug: Tigecycline

INTERVENTIONS:
Drug: Delafloxacin — Powder for solution for infusion 300 mg or tablet 450 mg, BID, for 5 to 14 days
  Arms: Delafloxacin
Drug: Vancomycin — Powder for solution for infusion 15mg/kg, BID, for 5 to 14 days
  Arms: Best Available Therapy
Drug: Linezolid — Solution for infusion or tablet, 600 mg BID, for 5 to 14 days
  Arms: Best Available Therapy
Drug: Piperacillin/Tazobactam — Powder for solution for infusion 4/0.5 g, TID, for 5 to 14 days
  Arms: Best Available Therapy
Drug: Tigecycline — Powder for solution for infusion 50 mg, TID, for 5 to 14 days
  Arms: Best Available Therapy

SUMMARY:
The purpose of this study is to assess the efficacy and safety of delafloxacin administered as IV and oral formulation in comparison with Best Available Therapy (BAT) in patients with superficial or deep incisional surgical site infection following a cardiothoracic/related leg or abdominal surgery.

DETAILED DESCRIPTION:
This is a randomized, observer-blinded, active-controlled, parallel-group, multicenter, phase IIIb study for the treatment of incisional, superficial or deep, surgical site infection after cardiothoracic /related leg or abdominal surgery (i.e patients who are at risk of microbiologically resistant infections). IV to be switched to oral delafloxacin will be compared to treatments that represent the best available therapy (BAT) for either cardiothoracic/related leg or abdominal surgical site infection (SSI).

Approximately 600 male and female eligible patients will be randomly assigned in a 1:1 ratio to receive delafloxacin or BAT. For patients who are randomised to BAT, the investigator will choose one out of two treatments available (two available for the cardiothoracic/related leg and two available for abdominal SSI) as most appropriate for patient characteristics and local epidemiological pattern.

Duration of study depends on treatment duration (range: minimum 5 to maximum 14 days, as per Investigator's judgment) followed by visits up to 30 days after end of treatment.

Patients will be hospitalized from Screening (within 30 days from surgery) and will remain hospitalized until considered improved or cure as per Investigator's judgment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged more than 18 years.
* Patients with a history of cardiothoracic / related leg or abdominal surgery, occurred within 30 days and no implant is left in place, and a diagnosis of superficial or deep SSI according to the CDC definition.
* The severity of infection requires an IV treatment and patient hospitalization according to the Investigator's judgment.

Exclusion Criteria:

* Previous IV antimicrobial therapy exceeding 24-hour duration during 72 hours prior to first dose.
* Any infection expected to require systemic antimicrobial agents other than study treatment(s).
* Medical history of significant hypersensitivity or allergic reaction or contraindication to the study drugs
* Medical history of central nervous system (CNS) disorders
* Medical history of myasthenia gravis.
* Medical history of C. difficile diarrhea.
* Organ-space infection.
* Complicated Intra-Abdominal Infection (cIAI)
* Chronic or underlying conditions at site of infection that may complicate the assessment of clinical response or would interfere with SSI healing.
* Underlying disease leading to deep immunosuppressive status.
* End-stage renal disease, CrCl <15 mL/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Margaritora, Principal Investigator — Hospital Agostino Gemelli
Locations (1):
- Hospital Agostino Gemelli, Roma, Italy

REFERENCES:
- [Derived] Belev N, Tein A, Mangialardi G, Nuti A, Marino Merlo G, Scartoni S, Bertolotti M, Lerro M, Margaritora S. A Randomized, Observer-Blinded, Active-Controlled, Phase IIIb Study to Compare IV/Oral Delafloxacin Fixed-Dose Monotherapy With Best Available Treatments in a Microbiologically Enriched Population With Surgical Site Infections: The DRESS Study. Open Forum Infect Dis. 2025 Aug 29;12(9):ofaf476. doi: 10.1093/ofid/ofaf476. eCollection 2025 Sep. PMID 40908975

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, the recruiment period lasted 13 months, since August 2019 to September 2020. The recruitment was mostly conducted at Abdominal and General surgery departments.
Pre-assignment Details: In total, 274 patients were screened while 266 patients were randomized and treated (ITT population).
Groups:
- Best Available Therapy: Cardiothoracic / related leg SSI
  * Vancomycin IV
  * Linezolid IV, with the option to switch to linezolid oral.
  In case of suspicion of Gram-negative, additional therapy shall be added as per investigator's choice
  Abdominal SSI
  * Piperacillin/Tazobactam IV, OR
  * Tigecycline IV
  In case of suspicion of MRSA, if the pre-selected treatment is Piperacillin/Tazobactam, additional therapy shall be added as per investigator's choice.
  Vancomycin: Powder for solution for infusion 15mg/kg, BID, for 5 to 14 days
  Linezolid: Solution for infusion or tablet, 600 mg BID, for 5 to 14 days
  Piperacillin/Tazobactam: Powder for solution for infusion 4/0.5 g, TID, for 5 to 14 days
  Tigecycline: Powder for solution for infusion 50 mg, TID, for 5 to 14 days
Period: Overall Study
Arm/Group | Delafloxacin | Best Available Therapy
Started | 134 | 132
Vancomycin IV | 0 | 2
Linezolid IV, With the Option to Switch to Linezolid Oral | 0 | 8
Piperacillin/Tazobactam IV | 0 | 68
Tigecycline IV | 0 | 54
Completed | 127 | 127
Not Completed | 7 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Death | 2 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT analysis population used as reference
Groups:
- Delafloxacin: Delafloxacin IV with the option to switch to OS
- Best Available Therapy: Vancomycin and Linezolid for cardiothoracic SSI Piperacillin/Tazobactam and Tigecycline for abdominal SSI
- Total: Total of all reporting groups
Arm/Group | Delafloxacin | Best Available Therapy | Total
Number analyzed (Participants) | 134 | 132 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (13.65) | 63.7 (13.71) | 64.9 (13.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 53 | 114
  Male | 73 | 79 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 131 | 131 | 262
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 133 | 132 | 265
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Site of infection [Count of Participants; unit: Participants]
  Abdominal SSI | 124 | 122 | 246
  Cardiothoracic SSI | 10 | 10 | 20
Depth of infection [Count of Participants; unit: Participants] — Superficial SSI, involving only skin and subcutaneous tissue of the incision, and at least one of the AND the patient has at least one of the infection symtomps
  * pain or tenderness,
  * localized swelling,
  * redness or heat;
  Or
  Deep SSI, involving deep soft tissues (e.g. fascia and muscle layers) at the incision site and at least one of the signs or symptoms of infection:
  * fever (> 38 °C),
  * localized pain or tenderness
  Participants
    Superficial SSI | 82 | 79 | 161
    Deep SSI | 52 | 53 | 105

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Success at Test Of Cure Visit
Description: Clinical Success defined as the clinical response of "Cure" or "improved". Below the definitions:
  * Cure: The complete resolution of all baseline signs and symptoms of SSI
  * Improved: two or more signs and/or symptoms (but not all) were considered resolved thus the patient had improved to an extent that no additional antibiotic treatment was necessary.
Time Frame: 7-14 days after last dose
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Best Available Therapy
Number analyzed (Participants) | 134 | 132
Participants | 123 | 119

2. Secondary Outcome: Hospital Infection Related Length of Stay (IRLOS)
Description: Length of Stay since beginning of therapy till patient stabilization and considered suitable for hospital discharge
Time Frame: up to 14 days
Population: CE population
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Delafloxacin: Delafloxacin IV with the option to switch to delafloxacin OS
Arm/Group | Delafloxacin | Best Available Therapy
Number analyzed (Participants) | 128 | 127
hours | 130.9 (71.87) | 140.3 (68.98)

3. Secondary Outcome: Hospital Length of Stay (LOS)
Description: Length of Stay since Screening till actual hospital discharge
Time Frame: up to 45 days (Late Follow Up visit)
Population: ITT population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Delafloxacin | Best Available Therapy
Number analyzed (Participants) | 134 | 132
hours | 178.8 (95.44) | 193.5 (119.72)

4. Secondary Outcome: Number of Participants Eligible to Switch to Oral Formulation According to Blinded Observer's Assessment
Description: Blinded assessment based on patient stabilization and ability to tolerate OS diet. In particular, the following details had to be met:
  Systolic blood pressure normal/not clinically significant abnormal No infection related tachycardia Afebrile status; body temperature <38°C for at least 24 hours* WBC count normalized/not clinically significant abnormal Patient able to tolerate PO diet/to take PO treatment and no GI absorption problem
  The measure counts only the participants eligible to switch, without taking into account the actually switched. Indeed, only linezolid in the BAT has an equivalent oral formulation suitable for the switch.
Time Frame: up to 14 days
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Best Available Therapy
Number analyzed (Participants) | 134 | 132
Participants | 129 | 129

5. Secondary Outcome: Microbiological Response
Description: Documented or presumed eradication or persistence
Time Frame: up to 14 days (End Of Treatment visit) and 7-14 days after last dose (Test Of Cure visit)
Population: MITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Best Available Therapy
Number analyzed (Participants) | 105 | 102
Participants
  TOC Visit: Eradicated | 94 | 81
  TOC Visit: Persisted | 11 | 21
  EOT Visit: Eradicated | 80 | 64
  EOT Visit: Persisted | 25 | 38

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant from the time of ICF signature (Screening) up to to LPLV, i.e. for maximum 45 days.
Groups:
- Best Available Therapy: Vancomycin and Linezolid for cardiothoracic SSI Piperacillin/Tazobactam and Tigecycline for abdominal SSI
  The results are not reported "per intervention" since the study was not powered to highlight difference between delafloxacin and each reference treatment. The safety analysis aimed to demonstrate that delafloxacin, among the fluoroquinolone class, is atypical showing a favourable safety profile very similar to NON-fluoroquinoles.
- Linezolid: Linezolid IV with the option to switch to delafloxacin OS
- Vancomycin: Vancomycin IV
- Piperacillin/Tazobactam: Piperacillin/Tazobactam IV
- Tigecycline: Tigecycline IV
Arm/Group | Delafloxacin | Best Available Therapy | Linezolid | Vancomycin | Piperacillin/Tazobactam | Tigecycline
All-Cause Mortality (participants affected / at risk) | 4/134 | 1/132 | 0/8 | 0/2 | 0/68 | 1/54
Serious Adverse Events (participants affected / at risk) | 9/134 | 14/132 | 1/8 | 0/2 | 10/68 | 3/54
Other Adverse Events (participants affected / at risk) | 22/134 | 26/132 | 2/8 | 0/2 | 18/68 | 6/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delafloxacin (N=134) | Best Available Therapy (N=132) | Linezolid (N=8) | Vancomycin (N=2) | Piperacillin/Tazobactam (N=68) | Tigecycline (N=54)
angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ileus (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
gas gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
postoperative wound complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delafloxacin (N=134) | Best Available Therapy (N=132) | Linezolid (N=8) | Vancomycin (N=2) | Piperacillin/Tazobactam (N=68) | Tigecycline (N=54)
diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pyrexia (General disorders) | 2 (2) | 1 (5) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Hypokalaemia (Investigations) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
hypophosphataemia (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
phlebitis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
anemia folate deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
anemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
thyroid mass (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
pancreatic calcification (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
post-operative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hypomagnaesemia (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT04042077/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT04042077/SAP_001.pdf